CLINICAL TRIAL: NCT01183754
Title: Use of a Point-of-Care Platelet Function Assay to Improve the Prediction of Atherothrombotic Events After Implantation of Drug-Eluting Stents: ASAN-VerifyNow Registry
Brief Title: Use of a Point-of-Care Platelet Function Assay for the Prediction of Atherothrombotic Events
Acronym: ASAN-VERIFY
Status: Completed | Type: Observational
Sponsor: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Clinical Research Center, Asan Medical Center
Other Study IDs: 200603
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2006-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; platelet reactivity; drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling for genotyping (genetic subgroup analysis)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients receiving drug-eluting stents

SUMMARY:
1. To evaluate the role of VerifyNow test as prognostic marker in routine clinical practice using drug-eluting stents.
2. To determine the add-on-effect of VerifyNow test beyond on conventional risk factors (clinical, lesions, or procedural factors).
3. To compare the prognostic utility of VerifyNow test with several biomarkers.

DETAILED DESCRIPTION:
Predictive role of a point-of-care assay (VerifyNow test) has not been well evaluated in large number of patients receiving drug-eluting stents as a routine practice.

In addition, additional predictive effect of a point-of-care assay, as compared to conventional clinical factors or other biomarkers, might be clinically interesting and important.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with established coronary artery disease receiving PCI with stent implantation

Exclusion Criteria:

* Cardiogenic shock
* Patients using concomitant medication known to affect platelet function other than aspirin (i.e. nonsteroidal antiinflammatory agents, dipyramidole, upstream glycoprotein IIb/IIIa inhibitors)
* patients with a known platelet function disorder or a whole blood platelet count of less than 150000/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included consecutive patients with de novo coronary artery disease who underwent an initial PCI with drug-eluting stents and had VerifyNow test at the Asan Medical Center (Seoul, Korea)
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2006-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause death, myocardial infarction, stent thrombosis, and stroke | at median 2 year after enrollment

SECONDARY OUTCOMES:
death (all-cause and cardiovascular) | at median 2 year after enrollment
myocardial infarction | at median 2 year after enrollment
stent thrombosis | at median 2 year after enrollment
stroke | at median 2 year after enrollment
Thrombolysis In Myocardial Infarction (TIMI) major/minor bleeding | at median 2 year after enrollment
target-vessel revascularization | at median 2 year after enrollment
Composite of cardiovascular death, MI, stent thrombosis, or stroke | at median 2 year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea